CLINICAL TRIAL: NCT03319186
Title: Pre-EDIT: A Randomised, Feasibility Trial of Elastance-Directed Intra-pleural Catheter or Talc Pleurodesis (EDIT) in the Management of Symptomatic Malignant Pleural Effusion Without Obvious Non-expansile Lung
Brief Title: EDIT Management Feasibility Trial
Acronym: Pre-EDIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Rocket Medical plc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN17ON084
Record Dates: First submitted 2017-08-04; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Pleural Effusion, Malignant
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Chest Tubes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EDIT Management (Experimental)
  Interventions: Procedure: EDIT Management
- Standard Care (Active Comparator)
  Interventions: Procedure: Chest drain and talc pleurodesis

INTERVENTIONS:
Procedure: EDIT Management — EDIT management
  1. Volumetric Pleural MRI for pre-aspiration pleural cavity volume
  2. Large volume pleural aspiration with recording of intra-pleural pressure during aspiration
  3. Volumetric Pleural MRI for post-aspiration pleural cavity volume
  4. Computation of PEL250, defined as the rolling average of pleural elastance over the preceding 250ml aspirated.
     MaxPEL250 ≥ 14.5 cm H2O/L: allocated to 1st-line IPC MaxPEL250 < 14.5 cm H2O/L: allocated to 1st-line TP
  5. EDIT-directed 1st-line treatment to be delivered within 24 hours; if insufficient residual pleural fluid to allow standard Seldinger insertion technique then Boutin-type needle used for pneumothorax induction and guide wire insertion.
  Arms: EDIT Management
Procedure: Chest drain and talc pleurodesis — Intercostal chest drain insertion and talc slurry instillation according to British Thoracic Society guidelines
  Arms: Standard Care

SUMMARY:
Malignant Pleural Effusion (MPE) is a collection of fluid inside the chest caused by cancer. It is a common medical problem and often causes severe breathlessness. Patients with this condition generally have a very poor survival and so it is extremely important that they are given effective treatment as soon as possible to minimise the amount of time they have to spend in hospital.

Standard treatment for MPE involves an admission to hospital to drain the fluid and then attempt to prevent the fluid from returning by sticking the lung to the inside of the rib cage with medical talc powder which acts like glue. This is called talc pleurodesis (TP) but unfortunately it fails in about 30% of patients. This is usually because the lung has not fully re-expanded and has not made contact with the inside of the ribs. When this happens, the fluid can be effectively treated with a different type of drainage tube called an indwelling pleural catheter (IPC) which tunnels under the skin and is drained at home by the district nurses.

It is thought that pressure measurements taken from the fluid as it is drained may be able to show doctors whether or not the lung will re-expand before patients are committed to either TP or an IPC. In this research we wish to test if these measurements can be used to choose which is the best first treatment option (TP or IPC) for patients with MPE. We have called this 'EDIT management'. Since it is uncertain whether this new approach will work, patients will be randomised to have either standard treatment or EDIT management. We will compare the two groups to assess whether the patients who had EDIT management had to have fewer repeat procedures over the following 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confident diagnosis of malignant pleural effusion, defined as any of the following:

  1. Pleural effusion with histocytologically proven pleural malignancy OR
  2. Pleural effusion in the context of histocytologically proven malignancy elsewhere, without a clear alternative cause for fluid OR
  3. Pleural effusion with typical features of malignancy with pleural involvement on cross-sectional imaging (CT/MRI)
* Degree of breathlessness for which therapeutic pleural intervention would be offered
* Age >18 years
* Expected survival > 3 months
* Written Informed Consent

Exclusion Criteria:

* Females who are pregnant or lactating
* Clinical suspicion of non-expansile lung for which talc pleurodesis would not be offered
* Patient preference for 1st-line indwelling pleural catheter (IPC) insertion
* Previous ipsilateral failed talc pleurodesis
* Estimated pleural fluid volume ≤ 1 litre, as defined by thoracic ultrasound
* Any contraindication to chest drain or IPC insertion, including:

Irreversible coagulopathy Inaccessible pleural collection, including lack of suitable IPC tunnel site

- Any contraindication to MRI scanning, including:

Claustrophobia Cardiac pacemaker Ferrous metal implants or retained ferrous metal foreign body Previously documented reaction to Gadolinium-containing intravenous contrast agent Significant renal impairment (eGFR<30 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruiting 30 patients within 12 months and randomising them to either EDIT Management or Standard Care | 12 months
  The number of patients recruited and randomised within 12 months

SECONDARY OUTCOMES:
Failure rate of the manometry procedure | 12 months
  Defined as the proportion of patients in whom PEL cannot be computed
Incidence of adverse events associated with the manometry procedure | 12 months
  Number of participants with Adverse Events (AEs) and Serious AEs (SAEs), defined by United Kingdom Good Clinical Practice in Research, associated with use of the digital pleural manometer
Aspiration threshold to detect abnormal pleural elastance | 12 months
  The pleural fluid aspiration volume at which the rolling average pleural elastance over the preceding 250ml (PEL250) first exceeds the upper limit of normal (14.5cm H2O/L).
Proportion of patients requiring pneumothorax induction following manometry | 12 months
  The proportion of patients in which pneumothorax induction is required to facilitate safe intercostal chest drain/IPC insertion in the EDIT arm (Group A)
Assess accuracy of pleural cavity volume change assumptions | 12 months
  To test the assumption that pleural cavity volume change is equivalent to the volume of pleural fluid removed during aspiration by measuring:
  1. Pleural fluid aspiration volume
  2. Pleural cavity volume change, as measured directly using volumetric Magnetic Resonance Imaging (MRI), calculated as pre- minus post-aspiration pleural cavity volume
Assess accuracy of ultrasound effusion volume estimate | 12 months
  To test the accuracy of a predictive model of pleural effusion volume based on thoracic ultrasound measurements by measuring:
  1. Thoracic ultrasound estimated total pleural effusion volume
  2. Pre-pleural fluid aspiration pleural cavity volume measured by volumetric MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Elizabeth University Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martin GA, Tsim S, Kidd AC, Foster JE, McLoone P, Chalmers A, Blyth KG. Pre-EDIT: A Randomized Feasibility Trial of Elastance-Directed Intrapleural Catheter or Talc Pleurodesis in Malignant Pleural Effusion. Chest. 2019 Dec;156(6):1204-1213. doi: 10.1016/j.chest.2019.07.010. Epub 2019 Jul 30. PMID 31374208
- [Derived] Martin GA, Tsim S, Kidd AC, Foster JE, McLoone P, Chalmers A, Blyth KG. Pre-EDIT: protocol for a randomised feasibility trial of elastance-directed intrapleural catheter or talc pleurodesis (EDIT) in malignant pleural effusion. BMJ Open Respir Res. 2018 May 29;5(1):e000293. doi: 10.1136/bmjresp-2018-000293. eCollection 2018. PMID 29862030